CLINICAL TRIAL: NCT01668394
Title: Effect of Learning and Coping Strategies in Cardiac Rehabilitation - A Randomised Controlled Parallel Group Study
Brief Title: Effect of Learning and Coping Strategies in Cardiac Rehabilitation - Group Study
Acronym: LC-REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Lynggaard, MHsc, PhD student at Cardiovasculat Research Unit, Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ethics app. number: 20100230
Record Dates: First submitted 2012-08-10; First posted 2012-08-20 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Rehabilitation
MeSH Terms: interventions — Educational Status; Coping Skills; Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Learning and coping arm (Active Comparator): Participation of experienced patients as co-educators. Completion of two individual clarifying interviews. Teaching style: situated, reflective, inductive.
  Interventions: Behavioral: Learning and coping arm
- Control arm (Placebo Comparator): Usual care. Teaching style: deductive.
  Interventions: Other: Control arm

INTERVENTIONS:
Behavioral: Learning and coping arm — Participation of experienced patients as co-educators. Completion of two individual clarifying interviews. Teaching style: situated, reflective, inductive.
  Other Names: Learning and coping strategies in cardiac rehabilitation
  Arms: Learning and coping arm
Other: Control arm — Usual care. Teaching style: deductive.
  Other Names: Standard cardiac rehabilitation
  Arms: Control arm

SUMMARY:
Background: It is well known that cardiac rehabilitation has potential to reduce morbidity and mortality, but not all patients complete CR. This LC-REHAB trial aims to compare the effect of a new patient education method called learning and coping strategies to that of standard care.

Design: Randomised controlled trial, 1:1 ratio. Participants: Patients above 18 years newly hospitalised with either ischaemic heart disease or heart failure.

Setting: Three hospital Units in Central Denmark Region. Intervention: Cardiac rehabilitation with addition of learning and coping strategies which include participation of experienced patients as co-educators, clarifuing interviews, and inductive teaching style.

Control arm: Standard care cardiac rehabilitation with a decuctive teaching style.

Outcomes: Adherence to cardiac rehabilitation, morbidity, mortality, risk factors, lifestyle, health related quality of life, return to work.

DETAILED DESCRIPTION:
Coronary heart disease is one the most common cause of death in Denmark and is also a chronic disease that 300,000 people in the country are living with. Cardiac rehabilitation is of great significance for this group of people because of its potential to reduce mortality and morbidity. However, not all patients succeed in changing their lifestyle in a positive and heart healthy direction. Thus, it is a great challenge to develop new methods which can help the patients to maintain a more healthy lifestyle in the long run. A concept for patient education, called learning and coping, has been developed in Norway. It is a health education method based on a high degree of involvement from the participants and on what is important for them. Planning, performance and evaluation happens in close cooperation between the health staff and so-called experienced patients. The course begins and ends with individual clarifying interviews.

The aim of this study is to evaluate the effect of learning and coping strategies in cardiac rehabilitation on adherence, risk factors and lifestyle, morbidity and mortality, health related quality of life and return to work.

The number of participants needed are estimated to 750 ptt.s with datacollection at baseline, just after rehabilitation, 3 months after rehabilitation and 3 years after rehabilitation. It is carried out as an open randomised controlled parallel group study in three hospitals in Hospital Unit West Jutland, Central Denmark Region, where the participants newly hospitalised with either ischemic heart disease or heart failure is randomised to either the intervention group with learning and coping strategies or to the standard group without the strategies. The rehabilitation courses in both groups last for eight weeks and consist of both training and education sessions. The concept of learning and coping is applied to the intervention group by letting 'experienced patients' participate in the education and not using standardised teaching slides. Also clarifying individual interviews are completed before and after the course. The 1:1 randomisation is computer generated and is stratified by hospital unit, diagnosis and gender. All analyses will be performed after the principle of 'intention to treat'.

The primary outcomes are adherence to cardiac rehabilitation, morbidity and mortality, while secondary outcomes are risk factors (blood pressure and lipid profile), lifestyle (body mass index, waist circumference, smoking status, exercise capacity and body compositions measured via DXA-scans) and health related quality of life (SF-12, Health Education Impact Questionnaire and Major Depression Inventory) and return to work (derived from the Danish Register for Evaluation of Marginalisation, (DREAM))

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years hospitalised with ichemic heart disease or heart failure motivated for completing a rehabilitation course

Exclusion Criteria:

* acute coronary syndrome less than five days before randomisation,
* active peri-, myo- or endocarditis,
* untreated symptomatic valvular disease,
* hypertension with systolic pressure over 200 mmHg and/or diastolic pressure over 110 mmHg,
* other extracardiac disease,
* planned revascularization,
* senile dementia,
* known compliance and former participation in the study.

Exclusion Criteria for outcome on return to work:

* age above 60 years
* recieving public transfer payments related to permanent work incapacity at week of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Adherence to cardiac rehabilitation | After 8 weeks of cardiac rehabilitation
Morbidity and mortality | Three or four years after last patient into trial

SECONDARY OUTCOMES:
Risk- and lifestyle factors | At baseline, after 8 weeks of rehabilitation, at 3 months after rehabilitation and at 3 years after rehabilitation
Health related Quality of life | At baseline, after 8 weeks of rehabilitation, at 3 months after rehabilitation and at 3 years after rehabilitation
Return to work | at baseline and after one year
  Four weeks of self support at follow up derived from the Danish Register for Evaluation of Marginalisation (DREAM)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Lynggaard, MHsc, Principal Investigator — Regional Hospital West Jutland
Locations (1):
- Regional Hospital West Jutland, Herning, Central Jutland, Denmark

REFERENCES:
- [Background] Lynggaard V, May O, Beauchamp A, Nielsen CV, Wittrup I. LC-REHAB: randomised trial assessing the effect of a new patient education method--learning and coping strategies--in cardiac rehabilitation. BMC Cardiovasc Disord. 2014 Dec 13;14:186. doi: 10.1186/1471-2261-14-186. PMID 25495543
- [Derived] Bitsch BL, Nielsen CV, Stapelfeldt CM, Lynggaard V. Effect of the patient education - Learning and Coping strategies - in cardiac rehabilitation on return to work at one year: a randomised controlled trial show (LC-REHAB). BMC Cardiovasc Disord. 2018 May 21;18(1):101. doi: 10.1186/s12872-018-0832-2. PMID 29783942
- [Derived] Lynggaard V, Nielsen CV, Zwisler AD, Taylor RS, May O. The patient education - Learning and Coping Strategies - improves adherence in cardiac rehabilitation (LC-REHAB): A randomised controlled trial. Int J Cardiol. 2017 Jun 1;236:65-70. doi: 10.1016/j.ijcard.2017.02.051. Epub 2017 Feb 21. PMID 28259552
- [Derived] Dehbarez NT, Lynggaard V, May O, Sogaard R. Learning and coping strategies versus standard education in cardiac rehabilitation: a cost-utility analysis alongside a randomised controlled trial. BMC Health Serv Res. 2015 Sep 28;15:422. doi: 10.1186/s12913-015-1072-0. PMID 26412226
- See also: BMC Cardiovascular Disorders — http://www.ncbi.nlm.nih.gov/pubmed/25495543